CLINICAL TRIAL: NCT00195767
Title: An Open-Label Long-Term Study to Evaluate the Safety of Depakote Extended Release Tablets in the Treatment of Mania Associated With Bipolar Disorder in Children and Adolescents
Brief Title: Evaluate the Safety of Depakote Extended Release Tablets in the Treatment of Mania Associated With Bipolar Disorder in Children and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M02-555
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2007-03-19 (Estimated); Status verified 2007-03

CONDITIONS: Bipolar I Disorder, Manic or Mixed
Keywords: Bipolar I Disorder; Depakote ER; divalproex sodium
MeSH Terms: conditions — Mania | interventions — Valproic Acid

INTERVENTIONS:
Drug: divalproex sodium

SUMMARY:
To determine if long-term treatment, up to 6 months, with Depakote ER is safe and effective in the treatment of bipolar I disorder in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Subject and subject's legal representative have voluntarily signed and dated an IRB-approved informed assent form and an IRB-approved informed consent form, respectively, before any study-specific procedures or tests are performed.
* The subject was randomized into Study M01-342 and either completed the study or prematurely discontinued due to ineffectiveness.
* The subject is male or a non-pregnant, non-lactating female.
* Subject is judged to be in general good health based upon the results of a physical examination, vital signs, 12-lead electrocardiogram (ECG), and laboratory profile (as described in Section 5.3.1)

Exclusion Criteria

* Subject is female, of childbearing potential, and not using an effective method of birth control (e.g., total sexual abstinence or contraceptives).
* Subject experienced a serious adverse event in Study M01-342, which the investigator considered "possibly" or "probably related" to study drug.
* Subject is violent, homicidal, or suicidal such that, in the opinion of the investigator, the subject is at significant imminent risk of hurting self or others.
* Subject has any of the following abnormal laboratory results at the last assessment prior to Day 1: Platelet count </= 100,000/µL; ALT or AST >/= 2 times Upper Limit of Normal (ULN)
* The subject is taking a protocol allowed medication for ADHD that has not been stable for at least 3 months prior to Day 1, is expected to require a dosage adjustment during the study, or that, in the investigators opinion, may be exacerbating mood symptoms.
* Subject requires treatment with or has taken a protocol-prohibited medication (see Appendix D) within 5 elimination half lives of Day 1.
* Subject has received an investigational drug, other than Depakote ER in Study M01-342, within 30 days prior to Day 1 of this study.
* In the investigator's opinion, long-term treatment with Depakote ER for the subject's mania associated with bipolar disorder is contraindicated.
* For any reason, subject is considered by the investigator to be an unsuitable candidate for this study.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150
Dates: Start 2004-07

PRIMARY OUTCOMES:
Safety outcome measures

SECONDARY OUTCOMES:
Y-MRS
CGI-S
C-GAS
CDRS-R
CGSQ
responders
remitters

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information 800-633-9110, Study Director — Abbott
Locations (1):
- Global Medical Information-Abbott, North Chicago, Illinois, United States

REFERENCES:
- [Derived] Wagner KD, Redden L, Kowatch RA, Wilens TE, Segal S, Chang K, Wozniak P, Vigna NV, Abi-Saab W, Saltarelli M. A double-blind, randomized, placebo-controlled trial of divalproex extended-release in the treatment of bipolar disorder in children and adolescents. J Am Acad Child Adolesc Psychiatry. 2009 May;48(5):519-532. doi: 10.1097/CHI.0b013e31819c55ec. PMID 19325497